CLINICAL TRIAL: NCT07020481
Title: Spiritual Needs of Patients With Inflammatory Bowel Disease and Their Caregivers: a European Cross-sectional Nursing Study
Brief Title: Spiritual Needs of European Patients With Inflammatory Bowel Disease and Their Caregivers
Acronym: Spirit@IBD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: SpNs-IBD-01
Record Dates: First submitted 2024-11-20; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A European-wide cross-sectional non-interventional study, initiated by a pilot study in Italy, will be conducted. The first phase of the pilot study is a 6-step translation, adaptation, and validation of the extended version of the Spiritual Needs Questionnaire (SpNQ-EV) and the Interpretation of Illness Questionnaire (IIQ) adopting the methodology [3] described in figure 1. To ensure they are both valid and user-friendly, the Thinking Out Loud (TOL) technique (think-aloud method) will pre-test their self-administration and provide fine tuning of the secondary objectives of the study. TOL involves participants verbalizing their thoughts while completing the questionnaires, allowing to capture real-time insights into their understanding, interpretation, and potential challenges with questionnaires' items. The second phase will consist of an anonymous e-survey consisting of the six questionnaires described in table 1 including the translated and validated SPNQ-EV and IIQ developed in phase 1. The European study will employ a multilingual anonymous e-survey developed to ensure accessibility in participants' native languages, eventually preceded by country-based pilot studies. Eligible participants include adolescents and adults with IBD, as well as their caregivers, recruited via nurses and patient associations.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and adults of all ages clinically diagnosed with CD, UC, or any other form of IBD (such as indeterminate colitis or IBD unclassified).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adults of all ages clinically diagnosed with CD, UC, or any other form of IBD (such as indeterminate colitis or IBD unclassified)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Spiritual Needs Questionnaire (SpNQ-EV) | Day 1 (From enrollment to the end of data collection (end of questionnaire completion) - same day
  To assess the spiritual needs among European IBD patients and their caregivers